CLINICAL TRIAL: NCT02826226
Title: Effect of Bronchodilatator Testing on Multiple-breath-washout (MBW) Derived Lung Function Parameters
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Dr. Frederik Trinkmann, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: MBW-bronchodilator
Record Dates: First submitted 2016-06-30; First posted 2016-07-07 (Estimated); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Obstructive Ventilation Disorders
MeSH Terms: interventions — Bronchodilator Agents

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- obstructive ventilation disorder: patients with known or suspected obstructive ventilation disorder and clinical indication for bronchodilator testing
  Interventions: Device: multiple-breath-washout test; Drug: Bronchodilator Agents

INTERVENTIONS:
Device: multiple-breath-washout test
Drug: Bronchodilator Agents

SUMMARY:
The investigators aim to evaluate the effect of bronchodilatator testing on multiple-breath-washout derived lung function parameters.

ELIGIBILITY:
Inclusion Criteria:

* known or suspected obstructive ventilation disorder
* clinical indication for bronchodilator testing

Exclusion Criteria:

* pregnancy
* inability to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with known or suspected obstructive ventilation disorder and clinical indication for bronchodilator testing
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
change of lung clearance index (LCI) as determined by multiple breath washout | 60 minutes

SECONDARY OUTCOMES:
repeatability of lung clearance index (LCI) | 60 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsmedizin Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No